CLINICAL TRIAL: NCT01976156
Title: The Gut-brain Axis: a Novel Target for Treating Behavioral Alterations in Obesity
Acronym: CIDO OEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 1308012537; 1R01CA180030 (NIH)
Record Dates: First submitted 2013-09-11; First posted 2013-11-05 (Estimated); Last update posted 2018-06-27 (Actual); Status verified 2018-06

CONDITIONS: Neural Response in Caudate; Weight Loss Trial; Impulsivity
MeSH Terms: conditions — Impulsive Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phopsholean dietary supplement (Experimental): Subjects in the Phospholean group will receive six capsules of PhosphoLean orally daily (total of 180 mg of NOPE and 120 mg of EGCG), ); two capsules consumed one hour before lunch, two capsules one hour prior to dinner, and two capsules two hours after dinner.
  Interventions: Dietary Supplement: PhosphoLean
- Placebo (rice flour) group (Placebo Comparator): The control (placebo) group will receive a placebo (identical in appearance, but containing 100 mg of rice flour per capsule).
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: PhosphoLean — PhosphoLean supplied by Cheminutra (White Bear Lake, MN). PhosphoLean® N-Oleoyl-PE + EGCG (NOPE + EGCG) is a proprietary phosphobioflavonic complex of N-oleoyl-phosphatidyl-ethanolamine (NOPE), which contains oleoyl ethanolamine (OEA) bound to phosphatidylethanolamine (PE), and epigallocatechin gallate (EGCG).
  Arms: Phopsholean dietary supplement
Dietary Supplement: Placebo — Placebo consists of rice flour
  Arms: Placebo (rice flour) group

SUMMARY:
The aims of this project are to determine if dietary supplementation with NOPE-EGCG (PhosphoLeantm, 30mg NOPE+20mg EGCG per capsule) can:

* rescue striatal function,
* increase adherence to a diet,
* reduce weight-gain after a diet,
* improve performance on impulsivity, go/no-go tasks, and negative outcome learning, and
* shift fat and sweet preference in overweight/obese human subjects

Secondary hypotheses: Baseline brain; perceptual and cognitive measures will be associated with diet, insulin sensitivity and may vary with genotype (TaqA1 1A polymorphism).

DETAILED DESCRIPTION:
In prior studies we have demonstrated an inverse relationship between body mass index and response in the dorsal striatum (DS) during consumption of a palatable milkshake (Stice et al. 2008). We have also shown that the magnitude of the reduced response predicts weight gain, especially in individuals who carry a copy of the A1 allele of the taq1A polymorphism (Stice et al. 2008). Since the A1 allele is associated with reduced striatal D2 receptors (Jonsson et al. 1999, Noble 2003, Noble et al. 1991, Pohjalainen et al. 1998, Ritchie et al. 1998, Thompson et al. 1997), this finding implicates the dopamine system in the reduced blood oxygen level dependent (BOLD) response. Our results also indicate that this reduced response is a consequence, rather than a cause of obesity, since gaining weight (Stice et al. 2010), but not risk for obesity (Stice et al. 2011) (by virtue of parental obesity), is associated with reduced DS response to palatable food. Taken together the results indicate that increased adiposity is associated with blunted DS response to palatable food that may reflect altered dopamine signaling. More recently we determined that reduced DS responses in overweight and obese subjects are associated with increased impulsivity measured with the Barratt Impulsiveness Scale and a go no/no-go task (Babbs et al, In Press).

Related to these findings in humans, preliminary work in rodents shows that exogenous administration of N-Acylethanolamines, such as oleoylethanolamine (OEA) can normalize high-fat diet induced dopamine decreases in DS and possibly induce a shift in preference (Tellez et al., In Press). Human testing of OEA supplementation is possible based on the availability of a dietary supplement containing the OEA precursor NOPE-EGCG ((PhosphoLEANtm, 100 mg NOPE+50mg EGCG per capsule). PhosphoLEAN has been shown to enhance adherence to dietary advice in overweight healthy subjects (Rondanelli et al. 2009, Mangine et al. 2012).

We therefore propose a double-blind cross-over study to test whether PhosphoLean will rescue striatal function, increase adherence to a diet, reduce weight-gain after a diet, improve performance on impulsivity, go/no-go tasks, and negative outcome learning, and shift fat and sweet preference in overweight/obese human subjects.

ELIGIBILITY:
Inclusion Criteria:

Right handed, English speaking, be a non-smoker (never smoked more than 2 cigarettes per month). Subjects will have a Body Mass Index > 25 kg/m2 (overweight/obese). Subjects are in good health. Subjects are able to provide a letter from their physician stating that they have had a physical exam in the past year and are in general good health and have specifically tested in the normal range for thyroid function and Hemoglobin 1Ac (and as such do not suffer from common metabolic disorders). In addition to this we will at intake confirm normal blood pressure, blood sugar and electrolyte balance for every subject.

Exclusion Criteria:

a) serious or unstable medical illness (e.g., cancer); b) past or current history of alcoholism or consistent drug use; c) current and history of major psychiatric illness as defined by the Diagnostic and Statistical Manual Diploma in Social Medicine-IV criteria including eating disorders, d) medications that affect alertness (e.g., barbiturates, benzodiazepines, chloral hydrate, haloperidol, lithium, carbamazepine, phenytoin, etc.)and any psychoactive drugs or anti-obesity agents; e) history of major head trauma with loss of consciousness; f) ongoing pregnancy; g) known taste or smell dysfunction; h) a diagnosis of diabetes; i) any known food allergy, certain food sensitivities (lactose); j) pregnant or nursing women, k) history of metalworking, injury with shrapnel or metal slivers, and major surgery; l) history of pacemaker or neurostimulator implantation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2013-10; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in neural response | 6 weeks, 5.5 months, 9.5 months
  change in neural response to milkshake stimulus will be measured with functional magnetic resonance imaging
Change in adherence to the behavioral weight loss program, greater weight loss maintenance,and these will be related to impulsivity, fat preference and intake, and striatal response | 5.5 months
  attendance to coaching sessions and food diaries will be used to measure adherence
Change in fat and sweet preference and intake | 6 weeks, 5.5 months, 9.5 months
  Subject will be asked to sample and rate fatty and sweet flavor stimuli (all made from commercially available ingredients).
Change in impulsivity | 6 weeks, 5.5 months, 9.5 months
  Various questionnaires and computer tasks addressing impulsivity

SECONDARY OUTCOMES:
Baseline brain | 0 weeks (baseline)
  perceptual and cognitive measures will be associated with diet, insulin sensitivity and may vary with genotype (TaqA1 1A polymorphism)

CONTACTS AND LOCATIONS:
Overall Officials: Dana M Small, PhD, Principal Investigator — The John B. Pierce Laboratory
Locations (1):
- The John B Pierce Laboratory, New Haven, Connecticut, United States

REFERENCES:
- [Background] Stice E, Spoor S, Bohon C, Small DM. Relation between obesity and blunted striatal response to food is moderated by TaqIA A1 allele. Science. 2008 Oct 17;322(5900):449-52. doi: 10.1126/science.1161550. PMID 18927395
- [Background] Jonsson EG, Nothen MM, Grunhage F, Farde L, Nakashima Y, Propping P, Sedvall GC. Polymorphisms in the dopamine D2 receptor gene and their relationships to striatal dopamine receptor density of healthy volunteers. Mol Psychiatry. 1999 May;4(3):290-6. doi: 10.1038/sj.mp.4000532. PMID 10395223
- [Background] Noble EP. D2 dopamine receptor gene in psychiatric and neurologic disorders and its phenotypes. Am J Med Genet B Neuropsychiatr Genet. 2003 Jan 1;116B(1):103-25. doi: 10.1002/ajmg.b.10005. PMID 12497624
- [Background] Noble EP, Blum K, Ritchie T, Montgomery A, Sheridan PJ. Allelic association of the D2 dopamine receptor gene with receptor-binding characteristics in alcoholism. Arch Gen Psychiatry. 1991 Jul;48(7):648-54. doi: 10.1001/archpsyc.1991.01810310066012. PMID 2069496
- [Background] Pohjalainen T, Rinne JO, Nagren K, Lehikoinen P, Anttila K, Syvalahti EK, Hietala J. The A1 allele of the human D2 dopamine receptor gene predicts low D2 receptor availability in healthy volunteers. Mol Psychiatry. 1998 May;3(3):256-60. doi: 10.1038/sj.mp.4000350. PMID 9672901
- [Background] Ritchie T, Noble EP. Association of seven polymorphisms of the D2 dopamine receptor gene with brain receptor-binding characteristics. Neurochem Res. 2003 Jan;28(1):73-82. doi: 10.1023/a:1021648128758. PMID 12587665
- [Background] Thompson J, Thomas N, Singleton A, Piggott M, Lloyd S, Perry EK, Morris CM, Perry RH, Ferrier IN, Court JA. D2 dopamine receptor gene (DRD2) Taq1 A polymorphism: reduced dopamine D2 receptor binding in the human striatum associated with the A1 allele. Pharmacogenetics. 1997 Dec;7(6):479-84. doi: 10.1097/00008571-199712000-00006. PMID 9429233
- [Background] Stice E, Yokum S, Blum K, Bohon C. Weight gain is associated with reduced striatal response to palatable food. J Neurosci. 2010 Sep 29;30(39):13105-9. doi: 10.1523/JNEUROSCI.2105-10.2010. PMID 20881128
- [Background] Stice E, Yokum S, Burger KS, Epstein LH, Small DM. Youth at risk for obesity show greater activation of striatal and somatosensory regions to food. J Neurosci. 2011 Mar 23;31(12):4360-6. doi: 10.1523/JNEUROSCI.6604-10.2011. PMID 21430137
- [Background] Rondanelli M, Opizzi A, Solerte SB, Trotti R, Klersy C, Cazzola R. Administration of a dietary supplement ( N-oleyl-phosphatidylethanolamine and epigallocatechin-3-gallate formula) enhances compliance with diet in healthy overweight subjects: a randomized controlled trial. Br J Nutr. 2009 Feb;101(3):457-64. doi: 10.1017/S0007114508024008. Epub 2008 Jul 1. PMID 18590587
- [Background] Mangine GT, Gonzalez AM, Wells AJ, McCormack WP, Fragala MS, Stout JR, Hoffman JR. The effect of a dietary supplement (N-oleyl-phosphatidyl-ethanolamine and epigallocatechin gallate) on dietary compliance and body fat loss in adults who are overweight: a double-blind, randomized control trial. Lipids Health Dis. 2012 Oct 4;11:127. doi: 10.1186/1476-511X-11-127. PMID 23033919